CLINICAL TRIAL: NCT04187495
Title: A Phase I Study for Tolerance and Pharmacokinetic Characteristic of MAX-40279 in Patients With Relapsed or Refractory Acute Myelogenous Leukemia
Brief Title: Study of MAX-40279 in Patients With Relapsed or Refractory Acute Myelogenous Leukemia (AML)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maxinovel Pty., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAX-40279-002
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: AML

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MAX-40279-01 (Experimental)
  Interventions: Drug: MAX-40279-01

INTERVENTIONS:
Drug: MAX-40279-01 — Part 1: Dose escalation, MAX-40279-01 twice daily with dose modifications based on tolerability criteria.
  Part 2: Dose expansion, Recommended doses from Part 1.
  For each dose level, a single dose of MAX-40279-01 will be first administered orally followed by 1 day observation, then continuous treatment will start 4 weeks treatment (per cycle).

SUMMARY:
This is a non-randomized, open-label, single-arm, dose-escalation Phase I study to evaluate the safety and tolerability of MAX-40279-01 in patients with Relapsed or Refractory AML.

DETAILED DESCRIPTION:
This is a two-part study comprised of a dose escalation part and a dose expansion part.

ELIGIBILITY:
Inclusion Criteria:

* Males and/or females over age 18.
* Subject has morphologically documented relapsed or refractoryprimary AML as defined by the World Health Organization (WHO) 2016 criteria for which no established standard therapy is available.
* ECOG performance status of 0 to 2.
* Persistent chronic clinically significant non-hematological toxicities from prior treatment (including chemotherapy, kinase inhibitors, immunotherapy, experimental agents, radiation, HSCT, or surgery) must be Grade ≤ 1.
* Any anti-tumor treatment with radiation therapy, surgery, or immunotherapy wihtin 2 weeks prior to trial entry.
* Life expectancy of at least 3 months.
* Both men and women of reproductive potential must agree to use a highly effective method of birth control during the study and for six months following the last dose of study drug.

Exclusion Criteria:

* Disease diagnosis of acute promyelocytic leukemia.
* Medical history of difficulty swallowing, malabsorption or other chronic gastrointestinal disease, or conditions that may hamper compliance and/or absorption of the tested product.
* Previously treated malignancies other than the current disease, except for adequately treated non-melanoma skin cancer, in situ cancer, or other cancer from which the subject has been disease-free for at least 5 years at the trial entry.
* Laboratory values not within the Protocol-defined range.
* Concomitant disease or condition that could interfere with the conduct of the trial, or that would, in the opinion of the Investigator, pose an unacceptable risk to the subject in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-04-16 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | 8 weeks
  Incidence of treatment-related AEs
Maximum tolerated dose (MTD） | 4 weeks
  MTD will be defined as the maximum dose level at which no more than 1 of 3 participants experience a dose-limiting toxicity (DLT) within the first 4 weeks of multiple dosing.
Phase II dose (RP2D) | 4 weeks
  The number and proportion of patients experiencing at least 1 dose-limiting toxicity (DLT) will be used as the primary measure to evaluate the RP2D of MAX-40279-01.

SECONDARY OUTCOMES:
Tmax | Approximately 4 weeks
  Time to maximum plasma concentration
Cmax | Approximately 4 weeks
  Maximum plasma drug concentration
AUC | Approximately 4 weeks
  Area under the time-concentration curve
t1/2 | Approximately 4 weeks
  Observed terminal half-life
Objective response rate (ORR) | 1 months (anticipated)
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on IRWG.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang, China